CLINICAL TRIAL: NCT01982877
Title: A Trial to Improve Surrogate Decision-Making for Critically Ill Older Adults
Brief Title: The Four Supports Study: Family Support Intervention in Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Douglas White, MD, MAS Vice Chair and Professor of Critical Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01AG045176-01 (NIH)
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Critically Ill Intensive Care Unit Patients; Physician-Family Communication in Intensive Care Units; Surrogate Decision-making for Critically Ill Patients
Keywords: decision making; values elicitation; patient centered care; Four Supports; Family Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Support Intervention (Experimental): Multifaceted family support intervention as well as ICU educational component.
  Interventions: Behavioral: Four Supports Intervention; Behavioral: Educational Control Intervention
- Educational Control (Experimental): ICU educational component
  Interventions: Behavioral: Educational Control Intervention

INTERVENTIONS:
Behavioral: Four Supports Intervention — The Four Supports Intervention is a multi-faceted intervention involving the addition of a trained nurse/social worker interventionist to the patient's care team who delivers four kinds of support: emotional support, communication support, decision support, and anticipatory grief support.
  Arms: Family Support Intervention
Behavioral: Educational Control Intervention — In addition to usual care, enrolled surrogates will receive two 15-minute education sessions about critical illness and mechanical ventilation on days 2 and 5, delivered by a research staff coordinator with education in critical care nursing.

SUMMARY:
The purpose of this study is to test the effectiveness of a multi-faceted communication intervention for family members of critically ill patients to reduce the family members' long-term symptoms of depression and anxiety.

DETAILED DESCRIPTION:
One in four elderly Americans die in or shortly after discharge from an intensive care unit. An expanding body of literature documents that physician-family communication and end-of-life care is poor in intensive care units. These deficiencies are associated with high rates of adverse psychological outcomes among surrogates, physician-family conflict, and life support decisions that may be inconsistent with patients' goals and preferences. There is a lack of information on practical, generalizable interventions that effectively improve this important aspect of care for elderly patients and their families.

The primary aim of this study is to evaluate the effectiveness of a multifaceted communication intervention as compared to an educational control to improve psychological outcomes among family members of critically ill patients, using a randomized, controlled trial design.

This randomized controlled trial involves adding a Family Support Specialist (FSS) to the clinical team to provide four types of support to the families of patients with advanced critical illness: emotional support, communication support (between the clinical team and the family), decisional support (education about the role of a surrogate decision maker) and anticipatory grief support.

The overall aim of the study is to improve the long-term psychological outcomes for family members of critically ill patients, to improve the quality of communication and decision-making between physicians and families, and to improve the patient-centeredness of care.

What happens in the study?

Patient is randomized to one of two groups:

1. INTERVENTION GROUP: Family Support Specialist is added to the clinical team to provide emotional support to the family and facilitate frequent communication with the clinical team.
2. CONTROL GROUP: Receives usual care with the addition of two educational sessions provided by the FSS to teach family members about the ICU environment.

What do participants need to do?

Family Members: Interact with the Family Support Specialist daily. Family Support Specialist addresses family needs and ensures that their questions are addressed.

Physicians: Collaborate with the Family Support Specialist to determine how best to support the family as well as attending clinician-family meetings.

Sample size: With a sample size of 300 patients (450 surrogates), the study is well powered to detect small and clinically important differences in the primary outcome measure Hospital Anxiety and Depression Score (HADS).The trial's original sample size of 400 patients (600 surrogates) was chosen to maximize the power to detect differences in a secondary outcome measure (costs) that required a substantially larger sample size than the primary outcome (HADS). Since the original power calculations were conducted, new data were published which indicated that cost analysis in this context will require an even larger sample size based one effect modification from whether the patient lived or died. Therefore, the Data and Safety Monitoring Board recommended revising the sample size to power the trial on the primary outcome (HADS), which required 300 patients (450 surrogates).

ELIGIBILITY:
Patient Inclusion criteria:

1. age ≥21,
2. lack of decision making capacity as determined by clinical examination by the attending physician,
3. APACHE II score ≥ 22, AND/OR
4. > 40% risk of death in hospital or >40% chance of severe long term functional impairment as judged by the patient's attending physician.

Patient Exclusion Criteria:

1. lack of a surrogate decision maker and
2. impending organ transplantation.
3. decisions regarding care and treatment already made
4. not currently participating in competing research study
5. Discharged prior to enrollment
6. Incarcerated.

Surrogate Inclusion criteria:

1. age ≥ 18 years,
2. self-identify as being involved in surrogate decision-making for the patient, up to a total of four family/surrogates.
3. able to give full informed consent, and
4. able to complete written questionnaires.

Surrogate Exclusion Criteria:

1. age <18 years old,
2. unable to read and understand English, and
3. unable to complete questionnaires due to physical or cognitive limitations.

Physician Inclusion criteria:

1) Eligible physicians will be the patient's primary attending or his/her designee. If an enrolled patient is cared for by more than one attending physician during their ICU stay, each will be consented.

Physician Exclusion Criteria:

1) Study investigators will be excluded as participants.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | participants will be followed six months following the patient's death or discharge from hospital, an expected average of 195 days
  Burden of anxiety and depression will be measured in family members 6 months after enrollment using the validated 14-item Hospital Anxiety and Depression scale (HADS).

SECONDARY OUTCOMES:
Patient and family-centeredness of care | At 6 months
  Patient and family-centeredness of care measured using the 12-item Patient-Perceived Patient-Centeredness of Care Scale (PPPC) adapted to use by surrogates.
Total Hospital Costs | Duration of hospital stay, an expected average of 4 weeks
  he costs are measured using aggregate data form the date of hospital admission through hospital discharge
Intensive Care Unit Length of Stay | Participants will be followed for duration of ICU stay, an expected average of 21 days
  The Intensive Care Unit length of stay , assessed by abstraction from hospital administrative records
Hospital Length of stay | Participants will be followed for duration of hospital stay, an expected average of 4 weeks
  Hospital length of stay length of stay , assessed by abstraction from hospital administrative records
Impact of Events scale at 6 months | at 6 months
  Symptoms of post traumatic stress in family members assessed using the validated 22 item Impact of Events Scale.

OTHER OUTCOMES:
Concordance between clinicians and surrogates about patient's prognosis (CSCS) | Participants are followed at time of enrollment, on day 5 of enrollment, and weekly thereafter for the duration of the hospital stay, an expected average of 4 weeks
  Prognostic estimates of survival and long-term functional impairment are measured responses by assessing the surrogate decision maker and the physician
Decisional Conflict Scale (DCS) | Participants are followed at time of enrollment and on day 5 of enrollment
  This validated instrument measures personal perceptions of:
  1. uncertainty in choosing options;
  2. modifiable factors contributing to uncertainty such as feeling uniformed, unclear about personal values and unsupported in decision making; and
  3. effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.
Quality of Communication Scale | Day 5 of enrollment
  Quality of communication in family members is assessed using the validated 19 item Quality of Communication Scale
Impact of Events Scale | at 3 months
  Symptoms of post traumatic stress in family members assessed using the validated 22 item Impact of Events Scale.
Inventory of Complicated Grief | At 3 months and at 6 months
  This validated instrument consists of 19 first-person statements concerning the immediate bereavement-related thoughts and behaviors of the participant.
Utilization of Mental Health Treatment | At 3 months and 6 months
  The utilization of mental health treatment is tracked via participant interview
Activity of Daily Living | At 6 months
  Functional status of the patient is assessed using the validated Katz Activities of Daily Living Scale.
Vital Status | At 6 months
  Mortality of the patient will be assessed at 6 months using hospital administrative records, and the 6-month follow-up with surrogate decision makers.
Discharge Dispensation | Participants will be followed for duration of hospital stay, an expected average of 4 weeks
  The disposition of the patient at time of discharge will be assessed via chart abstraction
HADS | at 3 months
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Butler RA, Seaman JB, Felman K, Stonehouse W, San Pedro R, Morse JQ, Chang CH, Lincoln T, Reynolds CF 3rd, Landefeld S, Happ MB, Song MK, Angus DC, Arnold RM, White DB. Randomized Clinical Trial of the Four Supports Intervention for Surrogate Decision-Makers in Intensive Care Units. Am J Respir Crit Care Med. 2025 Mar;211(3):370-380. doi: 10.1164/rccm.202405-0931OC. PMID 39586017
- [Derived] Seaman JB, Arnold RM, Buddadhumaruk P, Shields AM, Gustafson RM, Felman K, Newdick W, SanPedro R, Mackenzie S, Morse JQ, Chang CH, Happ MB, Song MK, Kahn JM, Reynolds CF 3rd, Angus DC, Landefeld S, White DB. Protocol and Fidelity Monitoring Plan for Four Supports. A Multicenter Trial of an Intervention to Support Surrogate Decision Makers in Intensive Care Units. Ann Am Thorac Soc. 2018 Sep;15(9):1083-1091. doi: 10.1513/AnnalsATS.201803-157SD. PMID 30088971